CLINICAL TRIAL: NCT02351622
Title: A Multicentre Randomized Study of Caffeic Acid Tablets as a Second-line Therapy for the Treatment of Immune Thrombocytopenia (ITP)
Brief Title: Caffeic Acid Tablets as a Second-line Therapy for ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Anhui Medical University (Other); Qingdao University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Caffeic acid
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — caffeic acid; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- caffeic acid tablet and dexamethasone (Experimental): Oral administration of caffeic acid tablet 0.3g three times per day for 1 year. Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later, 3 cycles in total.
  Interventions: Drug: Caffeic acid; Drug: Dexamethasone
- Placebo and dexamethasone (Active Comparator): Oral administration of placebo tablet 0.3g three times per day for 1 year. Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later, 3 cycles in total.
  Interventions: Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Caffeic acid — Oral administration of caffeic acid tablet 0.3g three times per day for 1 year
  Other Names: Caffeic acid tablet
  Arms: caffeic acid tablet and dexamethasone
Drug: Dexamethasone — Oral administration of dexamethasone 40 mg for four consecutive days then proceed another cycle 10 days later, 3 cycles in total.
Drug: Placebo — Sugar pills manufactured to mimic caffeic acid tablet. Oral administration of placebo tablet 0.3g three times per day for 1 year.
  Other Names: Placebo tablet
  Arms: Placebo and dexamethasone

SUMMARY:
The investigators are undertaking a multicentre, randomised controlled trial of 120 adults with newly diagnosed ITP from 5 medical centers in China. Part of the participants are randomly selected to receive caffeic acid tablets combining dexamethasone and the other part are selected to receive high-dose dexamethasone treatment. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

DETAILED DESCRIPTION:
All participants' platelet count will be monitored weekly. Response will be evaluated after 3, 6 and 12 months after treatment. If the participant did not get complete response or response after 3 months, he would quit the trail.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years
3. To show a platelet count <30 * 10^9/L, and with bleeding manifestations
4. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit
2. Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit
3. Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study
4. Current HIV infection or hepatitis B virus or hepatitis C virus infections
5. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test
8. Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proposed criteria for assessing response to ITP treatments | 3 months after treatment started
  1. Complete response (CR)： A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding.
  2. Response (R)： A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding.
  3. No response (NR)： A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.
  4. Relapses: platelet count falls below 30×10^9/L or bleeding accrues after achieving R or CR.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD, PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China